CLINICAL TRIAL: NCT00249717
Title: Group-Based Contingency Management for Substance Abuse Treatment
Brief Title: Group-Based Contingency Management for Substance Abuse Treatment - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-18883-1; R01DA018883 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Substance Abuse
Keywords: Contingency management; Substance abuse treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management — Receive rewards (prizes) abstinence and attendance

SUMMARY:
The purpose of this study is to evaluate the efficacy of prize-based contingency management (CM) when administered exclusively in groups. Substance dependent patients (N=360) at community-based treatment programs are randomly assigned to one of two conditions: (a) standard, non-CM treatment or (b) standard treatment plus prize CM delivered in groups. In the CM condition, patients earn the opportunity to win prizes for attending groups and submitting drug-free biological specimens. Substance use and psychosocial problems are measured at intake, month 1, month 3 (post treatment), and at 6-, 9-, and 12-month follow-up evaluations. We also assess patient characteristics that may be associated with improved outcomes within and across conditions.

ELIGIBILITY:
Inclusion criteria:

* age > 18 years
* current DSM-IV diagnosis of cocaine, opioid or alcohol abuse or dependence
* willing to provide breath and urine samples for 12 weeks
* English speaking
* willing to sign informed consent

Exclusion criteria:

* serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, severe or psychotic major depression, or suicide risk)
* dementia (<23 on the Mini Mental State Exam; Folstein et al. 1975)
* in recovery from pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2005-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Drug use | baseline and at each follow-up
Retention | each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States